CLINICAL TRIAL: NCT06575738
Title: Physiologic Response to Bariatric Surgery and the Impact of Adjunct Semaglutide - in Adolescents (the PRESSURE Trial)
Brief Title: Physiologic Response to Bariatric Surgery and the Impact of Adjunct Semaglutide in Adolescents
Acronym: PRESSURE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-3604; 5K23HL163480-02 (NIH)
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Adolescent Obesity; Body-Weight Trajectory; Weight Loss Trajectory; Bariatric Surgery; Anti-obesity Agents
Keywords: Obesity; Anti-obesity medication; Bariatric Surgery; Bariatric Surgery Post Operative Outcomes; Semaglutide; Sleeve gastrectomy
MeSH Terms: conditions — Obesity; Pediatric Obesity; Body-Weight Trajectory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Observational (No Intervention): Participants complete a set of standardized measures before bariatric surgery, 3 months postoperatively, and 12 months postoperatively.
- Active Medication + Standard Postoperative Care (Experimental): Participants can be enrolled between 1 and 2 years postoperatively and will receive usual interdisciplinary postoperative care plus weekly subcutaneous injectable semaglutide for 26 weeks. Initial dose is 0.25mg and is escalated every 4 weeks as tolerated (0.5mg, 1.0mg, 1.7mg, 2.4mg) for a total exposure of 26 weeks.
  Interventions: Drug: Injectable semaglutide; Behavioral: Standard postoperative care
- Standard Postoperative Care (Active Comparator): Participants can be enrolled between 1 and 2 years postoperatively and will receive usual interdisciplinary postoperative care.
  Interventions: Behavioral: Standard postoperative care

INTERVENTIONS:
Drug: Injectable semaglutide — Subcutaneous weekly injectable semaglutide
  Arms: Active Medication + Standard Postoperative Care
Behavioral: Standard postoperative care — Standard postoperative care consists of behaviorally-focused interventions delivered by the interdisciplinary Bariatric Surgery Center team targeting nutrition, physical activity, sleep, and mental health at standard postoperative intervals.
  Arms: Active Medication + Standard Postoperative Care; Standard Postoperative Care

SUMMARY:
The study plans to learn more about what happens to the body after bariatric surgery in people 12 to 24 years old. The study aims to understand why people respond differently to bariatric surgery and how to define success beyond weight loss alone. The study also plans to learn more about whether a medication (semaglutide) can help people 12 to 24 years old who, between 1 and 2 years after bariatric surgery, have not lost as much weight as expected.

ELIGIBILITY:
Observation Phase

Inclusion Criteria:

* Signed and dated informed consent form
* Willingness to comply with all study procedures and availability for the duration of the study
* Male or female biological sex, age 12 through 24 years
* In the preoperative pathway for vertical sleeve gastrectomy

Exclusion Criteria:

* Planned Roux-en-Y gastric bypass
* Hypothalamic obesity
* Type 2 Diabetes
* Current use of oral glucocorticoids (i.e. within 10 days of baseline visit)
* Current use of insulin

Intervention/Treatment Phase

Inclusion Criteria:

* Signed and dated informed consent form
* Status post vertical sleeve gastrectomy
* Male or female biological sex, age 12 through 24 years
* Meeting minimum nutrition goals
* Obesity: age 12-17 years: BMI ≥95th%ile for age/sex | age 18-24 years: BMI ≥ 30kg/m^2
* If entering the Intervention phase from the Observational phase: ≤20% BMI loss at 1 year postop
* If entering the Intervention phase from the existing patient pool: ≤20% BMI loss at 1-2 years postop

Exclusion Criteria:

* Surgically correctable cause of suboptimal postoperative weight loss
* Known hypersensitivity to any component of semaglutide
* Personal or family history of medullary thyroid carcinoma
* Personal history of multiple endocrine neoplasia type 2
* Hypothalamic Obesity
* Type 2 Diabetes
* History of pancreatitis
* Uncontrolled hypertension
* Clinically significant arrhythmia or heart disease that could be exacerbated by increased heart rate
* Malignant neoplasm within the last 5 years
* Untreated thyroid disorder
* Tanner Stage 1
* Baseline alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥ 5x upper limit of normal
* Baseline Creatinine >1.2mg/dL
* Active treatment for bulimia nervosa
* Active major psychiatric disorder limiting informed consent
* Suicidal ideation of type 4 or 5 on Columbia-Suicide Severity Rating Scale (C-SSRS)
* Intentional self-harm within the previous 1 month
* Severe unmanaged depression, defined by Center for Epidemiological Studies Depression (CESD) score of 26 or greater and by clinical evaluation
* Recent change to concomitant medications for hypertension, dyslipidemia, depression or anxiety (<4 weeks prior to enrollment)
* Use of oral glucocorticoids (within 10 days of baseline visit)
* Use of metformin (within 3 months of baseline visit)
* Use of insulin secretagogues (within 4 half-lives of the medication of baseline visit)
* Current use of insulin
* Use of anti-obesity medications (within 4 half-lives of the medication of baseline visit)
* Current pregnancy
* For females of reproductive potential: Plan to become pregnant in the next 8 months
* For females of reproductive potential: Not on contraception (i.e. two forms of birth control for example oral birth control pills and condoms) for at least 1 month prior to enrollment and agreement to use these during study participation and for an additional 8 weeks after the final dose of study medication

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Observational phase: Change in fasting glucagon-like peptide-1 (GLP1), measured by blood levels | Baseline, 12 months postoperatively
  GLP1 levels are measured prior to an oral mixed meal tolerance test
Observational phase: Change in stimulated glucagon-like peptide-1 (GLP1), measured by blood levels | Baseline, 12 months postoperatively
  GLP1 levels are measured during an oral mixed meal tolerance test
Observational phase: Change in insulin sensitivity (IS), measured by fasting blood insulin levels | Baseline, 12 months postoperatively
  Fasting insulin levels are measured. IS is defined as 1/fasting insulin
Observational phase: Change in percent fat free mass (FFM), measured by whole body dual-energy X-ray absorptiometry (DXA) | Baseline, 12 months postoperatively
  Percent FFM is calculated as (1-Percent Fat Mass) from DXA
Observational phase: Change in resting metabolic rate (RMR), measured by canopy indirect calorimetry | Baseline, 12 months postoperatively
  RMR from canopy indirect calorimetry
Observational phase: Change in 24 hour systolic blood pressure (BP), measured by ambulatory BP monitor | Baseline, 12 months postoperatively
  Mean 24 hour systolic BP
Observational phase: Change in indexed left ventricular mass (g/m to the 2.7th power), measured by echocardiogram | Baseline, 12 months postoperatively
  Resting supine 2-dimensional echocardiogram
Intervention phase: Change in BMI | Baseline, 26 weeks
  [(BMI at 26 weeks-Weight at Intervention Baseline)]/(BMI at Intervention Baseline)] * 100

SECONDARY OUTCOMES:
Change in fasting glucagon-like peptide-1 (GLP1), measured by blood levels | Baseline, 3 months postoperatively
  GLP1 levels are measured prior to an oral mixed meal tolerance test
Change in stimulated glucagon-like peptide-1 (GLP1), measured by blood levels | Baseline, 3 months postoperatively
  GLP1 levels are measured during an oral mixed meal tolerance test
Change in fasting Peptide YY (PYY), measured by blood levels | Baseline, 3 months postoperatively
  PYY levels are measured prior to an oral mixed meal tolerance test
Change in fasting Peptide YY (PYY), measured by blood levels | Baseline, 12 months postoperatively
  PYY levels are measured prior to an oral mixed meal tolerance test
Change in stimulated Peptide YY (PYY), measured by blood levels | Baseline, 3 months postoperatively
  Plasma PYY levels are measured during an oral mixed meal tolerance test
Change in stimulated Peptide YY (PYY), measured by blood levels | Baseline, 12 months postoperatively
  Plasma PYY levels are measured during an oral mixed meal tolerance test
Change in fasting ghrelin, measured by blood levels | Baseline, 3 months postoperatively
  Ghrelin levels are measured prior to an oral mixed meal tolerance test
Change in fasting ghrelin, measured by blood levels | Baseline, 12 months postoperatively
  Ghrelin levels are measured prior to an oral mixed meal tolerance test
Change in stimulated ghrelin, measured by blood levels | Baseline, 3 months postoperatively
  Ghrelin levels are measured during an oral mixed meal tolerance test
Change in stimulated ghrelin, measured by blood levels | Baseline, 12 months postoperatively
  Ghrelin levels are measured during an oral mixed meal tolerance test
Change in insulin sensitivity (IS), measured by fasting blood insulin levels | Baseline, 3 months postoperatively
  Fasting insulin levels are measured. IS is defined as 1/fasting insulin
Change in percent fat free mass (FFM), measured by whole body dual-energy X-ray absorptiometry (DXA) | Baseline, 3 months postoperatively
  Percent FFM is calculated as (1-Percent Fat Mass) from DXA
Change in resting metabolic rate (RMR), measured by canopy indirect calorimetry | Baseline, 3 months postoperatively
  RMR from canopy indirect calorimetry
Change in 24 hour systolic blood pressure (BP), measured by ambulatory BP monitor | Baseline, 3 months postoperatively
  Mean 24 hour systolic BP
Change in indexed left ventricular mass (g/m to the 2.7th power), measured by echocardiogram | Baseline, 3 months postoperatively
  Resting supine 2-dimensional echocardiogram
Intervention Phase: Eligibility rate | Up to 150 weeks
  (Patients meeting inclusion and exclusion criteria/Total patients screened)*100
Intervention Phase: Enrollment rate | Up to 154 weeks
  (Participants enrolled/Patients eligible)*100
Intervention Phase: Retention rate | Up to 184 weeks
  (Participants completing all intervention visits/Patients enrolled)*100
Intervention Phase: Mean maximum tolerated semaglutide dose | Baseline, 26 weeks
  Mean maximum tolerated dose (mg) of weekly injectable semaglutide
Intervention Phase: Number of participants with at least one serious adverse event (AE) in the active medication group, measured by a count | Up to 30 weeks
  Individual participants with serious AEs will be counted
Intervention Phase: Number of participants with an adverse event (AE) that leads to discontinuation of the medication, measured by a count | Up to 30 weeks
  Participants experiencing an AE that leads to medication discontinuation will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Moore, MD MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States